CLINICAL TRIAL: NCT07058675
Title: Myoinositol Therapy May Adjust The Metabolic Deregulation in Infertile Polycystic Ovarian Syndrome (PCOS) Women Through Modulation of The TyG Index-BMI: A Comparative Study Versus Metformin
Brief Title: Myoinositol vs. Metformin for Polycystic Ovarian Syndrome (PCOS): Impact on Metabolic Health and Fertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Basma Sakr, Assistant Professor of Obstetrics & Gynecology, Faculty of Medicine, Benha University, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC 1-11-2024
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: PCOS
MeSH Terms: interventions — Metformin; Inositol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myoinositol Group (Active Comparator): Patients presenting manifestations suggestive of having PCOS were evaluated for enrollment in the study, and took the tablets containing myoinositol/d-chiro-inositol combination (MYO/DCI) in 40:1 ratio
  Interventions: Drug: Myoinositol
- Metformin Group (Active Comparator): Patients presenting manifestations suggestive of having PCOS were evaluated for enrollment in the study, and took metformin (MET) hydrochloride 500 mg
  Interventions: Drug: Metformin Hydrochloride 500 MG

INTERVENTIONS:
Drug: Metformin Hydrochloride 500 MG — metformin (MET) hydrochloride 500 mg three times daily as the standard insulin sensitizer.
  Arms: Metformin Group
Drug: Myoinositol — myoinositol/d-chiro-inositol combination (MYO/DCI) in 40:1 ratiotwice daily
  Other Names: myoinositol/d-chiro-inositol combination (MYO/DCI) in 40:1 ratio
  Arms: Myoinositol Group

SUMMARY:
The study aimed to assess how a 6-month insulin sensitizer therapy impacts insulin resistance, glucose tolerance, and hormonal levels in women with PCOS. Researchers evaluated 156 PCOS patients, measuring their BMI, HOMA-IR (for insulin resistance), TyG index, TyG index-BMI, and total testosterone. Participants were divided into two groups, receiving either metformin or a myoinositol/d-chiro-inositol combination for six months, after which all parameters were re-evaluated to determine the percentage of change.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting manifestations suggestive of having PCOS;
* Patients were free of exclusion criteria.

Exclusion Criteria:

* Patients who were maintained on a diet regimen, or/and regular exercise;
* Patients who were on medical therapy of PCOS, antidiabetic or/and antihypertensive therapy;
* Patients who underwent laparoscopic drilling;
* Patients with dyslipidemia, hereditary lipoprotein disorders:
* Patients with chronic liver or kidney diseases.

Ages: 23 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Success Rate of Treatment Regimens in Restoring Menstrual Regularity and/or Achieving Pregnancy | 6~7 Months
  The proportion of patients who regained a regular menstrual pattern and/or achieved pregnancy during the study, reflecting the effectiveness of the administered treatment regimens.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha university, Banhā, El Qalyoubia, Egypt